CLINICAL TRIAL: NCT04581278
Title: Validation Study of the Feasibility of an Integrated Diagnostic System of Anatomo-pathological Lesions - Including Rejections - Appearing in Renal Grafts in the First Year of Transplant for Applicability in Routine Clinical Practice : KTD Innov-2 Study
Acronym: KTD Innov-2
Status: Completed | Type: Observational
Sponsor: Nantes University Hospital (Other)
Collaborators: Hôpital Necker-Enfants Malades (Other); Saint-Louis Hospital, Paris, France (Other)
Responsible Party: Sponsor
Other Study IDs: RC20_0284
Record Dates: First submitted 2020-09-03; First posted 2020-10-09 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Kidney Transplant
Keywords: Kidney Transplant; Integrated Diagnostic System

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — The blood, urine and biopsy samples required for the construction of the SDI will be completed upon inclusion in the KTD Innov-2 protocol (D0 of the graft, blood, urine) then at 3 months (monitoring biopsy of the renal graft, blood and urine) and 12 months (kidney transplant monitoring biopsy, blood and urine) in the 300 incident patients from the 3 university hospitals of the study (Nantes, Necker and Paris Saint-Louis). A blood and urine sample will accompany each graft biopsy which will be indicated in the first year of transplant.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: KTD Innov-2 — The main objective of the present study (KTD Innov-2) is to validate the feasibility of SDI within a limited time frame to ensure its clinically relevant use, with a high level of evidence to consider its labelling as a medical device by health authorities prior to routine transfer and/or future marketing.
  300 kidney transplant patients will be included in the KTD Innov-2 study with data collection, blood, urine and graft biopsies for biomarker analysis and conversion to SDI (decisional algorithms) and interactive multi-dimensional presentation on a web interface for use of the tool by transplant physicians and their patients.

SUMMARY:
The main objective of the present study (KTD Innov-2) is to validate the feasibility of SDI within a limited time frame to ensure its clinically relevant use, with a high level of evidence to consider its labelling as a medical device by health authorities prior to routine transfer and/or future marketing.

ELIGIBILITY:
Inclusion Criteria :

* Male and female patients, age ≥ 18 years at time of transplantation.
* Patients with a minimum weight of 40 kg in order to allow blood samples to be taken safely in accordance with the table published in the Order of 12 April 2018 setting the list of research mentioned in 3° of Article L. 1121-1 of the Public Health Code.
* Patients receiving a kidney transplant from a living or brain-dead donor.
* Patients expressing their non-opposition and ready to comply with the study procedures.

Exclusion Criteria :

* Patients who have received a previous transplant with an organ other than the kidney
* Patients unable or unwilling to perform study procedures or who do not speak French
* Vulnerable patients (minors, adults, pregnant women, under guardianship)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Inclusion of patients receiving a kidney transplant from a living donor Inclusion of patients receiving a kidney transplant from a deceased donor
  300 patients from 3 French centers routinely performing surveillance kidney graft biopsies at 3 months and 1 year of grafting. The 3 centres participating in the KTD Innov-2 study are the Nantes, Necker and Saint-Louis University Hospitals (Paris).
Sampling Method: Probability Sample
Enrollment: 210 (Actual)
Dates: Start 2021-06-02 (Actual); Primary Completion 2023-07-05 (Actual); Study Completion 2023-07-05 (Actual)

PRIMARY OUTCOMES:
Collection of biological samples necessary for the construction of the SDI | 12 months
  Validation of the circuit for the collection of the blood, urine and biopsy samples
Validation of the sample circuit from clinical unit to processing platforms | 12 months
  Path of the biological samples (blood, urine, biopsies) to the sample processing platforms for the editing of the raw results of the blood and urine and biopsy biomarkers
Validation of raw results transmission | 12 months
  The transmission of the raw results in the format necessary for the calculation of the diagnostic and/or prognostic algorithms
Validation of a final report | 12 months
  Edition of a final numerical report of the algorithms accessible on a web support with an intelligible interpretation by clinicians and patients.

SECONDARY OUTCOMES:
Validation of the diagnostic and/or prognostic capabilities of the SDI | 12 months
  The primary secondary endpoints will be to evaluate the sensitivity and specificity, as well as the negative and positive predictive values of the SDI obtained in the KTD innov-1 study, from an incident cohort of 300 new kidney transplant patients meeting the same inclusion criteria as the first KTD innov-1 study
Providing a final report of the SDI via web interfaces | 12 months
  The second secondary objective is to validate the integration of the algorithms in the SDI presentation software package

CONTACTS AND LOCATIONS:
Locations (1):
- Nantes University Hospital, Nantes, Loire-Atlantique, France

IPD SHARING:
Plan to Share IPD: Yes
eCRF
  The collection of data on each person suitable for research is carried out through a coded database. This coded database will be extracted from the existing DIVAT database in each participating centre, and the variables specific to the KTD Innov study (patient identification number (centre number/patient number) for the study, inclusion/non-inclusion criteria, date of collection of the non-opposition, additional analyses, ...) will be added on specific tabs.